CLINICAL TRIAL: NCT03605277
Title: A Phase I, Open-label and Single-dose Study to Evaluate the Pharmacokinetics and Safety of a Single 40 mg Oral Dose of ABL001 (Asciminib) in Subjects With Impaired Renal Function Compared to Matched Control Subjects With Normal Renal Function
Brief Title: Pharmacokinetics Study of Asciminib in Subjects With Impaired Renal Function Compared to Matched Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CABL001A2105; 2018-001394-25 (EudraCT Number)
Record Dates: First submitted 2018-07-20; First posted 2018-07-30 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Renal Impairment
Keywords: ABL001; asciminib; impaired renal function; pharmacokinetics
MeSH Terms: conditions — Renal Insufficiency | interventions — asciminib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Normal renal function (Experimental): healthy volunteers with normal renal function
  Interventions: Drug: Asciminib
- Severe renal impairment (Experimental): subjects with severe renal impairment
  Interventions: Drug: Asciminib
- Moderate renal impairment (Experimental): subject with moderate renal impairment
  Interventions: Drug: Asciminib
- Mild renal impairment (Experimental): subjects with mild renal impairment
  Interventions: Drug: Asciminib

INTERVENTIONS:
Drug: Asciminib — 40 mg single dose
  Other Names: ABL001

SUMMARY:
The purpose of this study is to characterize the pharmacokinetics (PK) and safety profile of asciminib following a single oral dose in adult subjects with renal impairment compared to a matched group of healthy subjects with normal renal function.

The results will determine whether or not a dose adjustment should be recommended when treating patients with asciminib who have impaired renal function.

ELIGIBILITY:
Inclusion Criteria:

* Male or sterile / post-menopausal female
* BMI between 18 and 36 kg/m2, body weight greater than or equal to 50 kg and no more than 120 kg
* Adequate venous access for blood sampling
* For healthy volunteers: subject must be matched to at least one renal impaired subject by age (+/- 10 years), body weight (+/- 20%) and gender
* For renal impaired subjects: documented stable renal disease without evidence of progressive decline in renal function (stable renal disease is defined as no significant change, such as, stable aGFR < 90, for 12 weeks prior to study entry)

Exclusion Criteria:

* women of child-bearing potential / pregnant / nursing
* contraindication or hypersensitivity to any drug or metabolites from similar class as asciminib or to any excipients of the study drug
* cardiac or cardiac repolarization abnormality
* history of psychiatric illness within the past 2 years
* history of acute or chronic pancreatitis
* subject on dialysis
* smokers (use of tobacco products in the previous 3 months) and not willing to abstain from using tobacco during the study
* any surgical or medical condition altering the absorption, distribution, metabolism or excretion of drug
* history of immunodeficiency diseases, including a positive Human Immunodeficiency Virus (HIV) test result at screening
* chronic infection with Hepatitis B virus (HBV) or Hepatitis C virus (HCV) at screening
* donation or loss of 400 mL or more of blood or plasma within 8 weeks prior to dosing or other amount considered to compromise the health of the subject if previous history of anemia exists
* use of the following drugs within 28 days prior to dosing: drugs that prolong the QT interval; CYP3A4 inhibitors and inducers; BCRP, UGT and PgP inhibitors and inducers

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-11-16 (Actual); Primary Completion 2019-03-18 (Actual); Study Completion 2019-04-14 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics: Plasma concentration of asciminib by AUClast | pre-dose (0 hour) and at 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48 and 72 hours post-dose
  The AUC from time zero to the last measurable concentration sampling time (tlast) (ng*h/mL)
Pharmacokinetics: Plasma concentration of asciminib by AUCinf | pre-dose (0 hour) and at 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48 and 72 hours post-dose
  The AUC from time zero to infinity (ng*h/mL)
Pharmacokinetics: Plasma concentration of asciminib by Cmax | pre-dose (0 hour) and at 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48 and 72 hours post-dose
  The maximum (peak) observed plasma, blood, serum, or other body fluid drug concentration after single dose administration (ng/mL)
Pharmacokinetics: Clearance of asciminib from plasma by CL/F | pre-dose (0 hour) and at 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48 and 72 hours post-dose
  The total body clearance of drug from the plasma (L/h)

SECONDARY OUTCOMES:
Asciminib PK parameters unbound AUClast (AUClast)u and unbound AUCinf (AUCinf)u based on unbound fraction in plasma | pre-dose (0 hour) and at 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48 and 72 hours post-dose
  including but not limited to: (AUClast)u: area under the unbound plasma concentration-time curve calculated to the last quantifiable concentration point (ng*h/mL)),
  - (AUCinf)u: unbound plasma concentration-time curve extrapolated to infinity. It is calculated as AUCinf ,u= AUClast ,u+ Clast,u/Lambda_z. (ng*h/mL)
Asciminib PK parameters unbound Cmax (Cmax)u based on unbound fraction in plasma | pre-dose (0 hour) and at 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48 and 72 hours post-dose
  The observed maximum unbound plasma concentration following administration (ng/mL)
Asciminib secondary PK parameters Tmax, T1/2 | pre-dose (0 hour) and at 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48 and 72 hours post-dose
  including but not limited to:
  * Tmax: the time to reach maximum (peak) plasma, blood, serum, or other body fluid drug concentration after single dose administration (h)
  * T1/2: the elimination half-life associated with the terminal slope (lz) of a semi logarithmic concentration-time curve (h).
Asciminib secondary PK parameter AUC0-72h | pre-dose (0 hour) and at 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48 and 72 hours post-dose
  The area under the unbound plasma concentration-time curve from time zero to 72 h post-dosing (ng*h/mL)
Asciminib secondary PK parameters Vz/F | pre-dose (0 hour) and at 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48 and 72 hours post-dose
  apparent unbound drug volume of distribution during the terminal elimination phase following extravascular administration
Percentage of participants with plasma protein binding as expressed by unbound fraction in plasma | 2 hours post-dose
  asciminib plasma protein binding in subjects with impaired renal function and subjects with normal renal function

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Novartis Investigative Site, Sofia, Bulgaria
- Novartis Investigative Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hoch M, Sato M, Zack J, Quinlan M, Sengupta T, Allepuz A, Aimone P, Hourcade-Potelleret F. Pharmacokinetics of Asciminib in Individuals With Hepatic or Renal Impairment. J Clin Pharmacol. 2021 Nov;61(11):1454-1465. doi: 10.1002/jcph.1926. Epub 2021 Jul 16. PMID 34115385
- See also: Results for CABL001A2105 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17610
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=616